CLINICAL TRIAL: NCT06312280
Title: Obiasity Study: Evaluation of Body Composition in Pediatric Patients With Overweight or Obesity
Brief Title: Evaluation of Body Composition in Pediatric Patients With Overweight or Obesity
Acronym: OBIASITY
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Simonetta Bellone, Professor, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: CE342/2023
Record Dates: First submitted 2024-02-12; First posted 2024-03-15 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Pediatric Obesity
Keywords: pediatric; obesity; overweight; body composition
MeSH Terms: conditions — Pediatric Obesity; Obesity; Overweight | interventions — Diet, Mediterranean

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric children and adolescents with obesity or overweight: The study will include all children and adolescents who visit the SCDU of Pediatrics, Surgery of Endocrinology and Auxology of the Major Charity Hospital of Novara for first visit or checkup for excess weight between 1 January 2024 and 30 May 2024 of both sexes that meet the following criteria of inclusion:
  Criteria for inclusion:
  Age between 6 and 17 years; BMI compatible with obesity or overweight according to IOTF criteria (6) Signature of informed consent by parents/legal guardians.
  Criteria for exclusion:
  Age below 6 years or over 18 Previous diagnosis of diabetes mellitus type 2 already placed in dietary or pharmacological therapy Subjects already included in dieto-therapeutic regimen Obesity secondary to diseases: genetic (Prader Willi syndrome, Down syndrome); metabolic and endocrine (Cushing syndrome, hypothyroidism)
  Interventions: Behavioral: Mediterranean diet

INTERVENTIONS:
Behavioral: Mediterranean diet — The composition of the diet will be distributed as follows: 55-60% of carbohydrates (45-50% complex carbohydrates and no more than 10% of simple sugars), 25-30% of lipids and 15% of proteins. It will be studied in accordance with the LARN (Italian Society of Human Nutrition, 2014) guidelines.

SUMMARY:
In recent decades, the prevalence of obesity and overweight has dramatically increased globally, representing a serious problem for society and for the health system of many countries, estimating an impact of 2-8% on global health spending. Obesity and overweight represent a problem not only for adults but also for children and adolescents: the latest data from the WHO estimate that about 340 million children and adolescents between 5 and 19 years are overweight or obese, data that increase drastically since 1975 from 4% of boys to 18% in 2016. (World Health Organization (WHO). The reduction and prevention of overweight and obesity in childhood is one of the main missions of public health at the global level, both for short-term and long-term implications. Recently, the importance of bioprothesiometric analysis (BIA) in the clinical routine has been evaluated, as it allows an estimation of body composition that would not otherwise be provided by the growth curves and the calculation of the Body Mass Index (BMI). In this study the investigators want to evaluate, in addition to the classic clinical parameters, the body composition of patients evaluated by means of an impedance balance (named TANITA MC780 MA P). With this study the investigators aim to investigate possible clinical and body composition changes in children and adolescents suffering from overweight and obesity with the ultimate aim of reducing cardio-metabolic risk factors related to it.

The objective of the study is the assessment of body composition, as an indicator of accuracy of lean mass, but especially of fat mass, of pediatric patients who are overweight and obesity in order to carry out a more complete evaluation of the clinical-metabolic condition for the prevention of cardiovascular risk.

The secondary objective is to assess the dietary compliance of the patients being studied and the possible correlation with the body composition.

DETAILED DESCRIPTION:
MATERIALS AND METHODS

The study will include all children and adolescents who visit the SCDU (Struttura Complessa a Direzione Universitaria) of Pediatrics, Surgery of Endocrinology and Auxology of the Major Charity Hospital of Novara for first visit or checkup for excess weight between 1 January 2024 and 30 May 2024 of both sexes that meet the following criteria of inclusion:

Criteria for inclusion:

Age between 6 and 17 years; BMI compatible with obesity or overweight according to International Obesity Task Force (IOTF) criteria Signature of informed consent by parents/legal guardians.

Criteria for exclusion:

Age below 6 years or over 18 Previous diagnosis of diabetes mellitus type 2 already placed in dietary or pharmacological therapy Subjects already included in dieto-therapeutic regimen Obesity secondary to diseases: genetic (Prader Willi syndrome, Down syndrome); metabolic and endocrine (Cushing syndrome, hypothyroidism)

Informed consent After reading the study fact sheet, patients will only be enrolled after the signature of the informed consent form by both parents or the legal representative and the minor subjects recruited (see patient and parent/guardian information attached to the protocol).

Upon enlistment (V1), the subjects included will undergo a clinical examination in accordance with normal practice, in which a bioimpedance analysis for the assessment of body composition is provided. The impedance analysis will be carried out using TANITA MC-780MA balance.

After the bioimpedance analysis and the clinical visit, a food scheme based on the Mediterranean Diet will be delivered. The composition of the diet will be distributed as follows: 55-60% of carbohydrates (45-50% complex carbohydrates and no more than 10% of simple sugars), 25-30% of lipids and 15% of proteins. It will be studied in accordance with the Reference Nutrient and Energy Intake Levels (LARN) (Italian Society of Human Nutrition, 2014) guidelines.

Follow-up Patients will be evaluated at the time of enrollment (V1), after 3 months (V3) and after 6 months (V6) as per clinical practice.

At the recruitment visit (V1) the following demographic and medical history of the patient and family will be collected:

sex, gender, age (years), ethnicity, weight and length at birth, type and duration of breastfeeding, age of parents (years), family history of previous diseases (Arterial Hypertension, Dyslipidemia, Hepatic Steatosis, Diabetes (specify if type I or II and oral or insulin therapy) and cardiovascular pathology, the smoking habit of parents, presence of gestational maternal diabetes), socioeconomic level of the family nucleus.

At all times (V1,V3,V6) the following assessments will be made:

Anthropometric measurements Height Weight BMI and BMI standard deviation score (SDS) Growth percentile according to Cacciari curves Waist/hips circumference, waist/height ratio Bioimpedance Pa and heart rate Stadium of Tanner Eating habits and medical history Semi-quantitative food frequency questionnaire (24h recall) Questionnaire of adherence to the Mediterranean diet called Quality Index for Children and Adolescents (KIDMED) Questionnaire on daily physical activity (IPAQ)

Biochemical assessments will also be carried out at the beginning and end of the protocol (V1 and V6) according to normal clinical practice (basic blood chemistry and/or OGTT). The analysis will be carried out at the clinical biochemistry laboratory of the University hospital (AOU- Azienda Ospedaliero Universitaria) "Major of Charity" of Novara.

During the biochemical evaluations, two serum and two plasma samples will be taken for Asprosin, Irisin and Ghrelin for the research of new markers related to obesity and its complications. The analysis will be carried out at the Laboratory of Biochemistry of the University of Eastern Piedmont The determination of clinical parameters will be carried out locally at the clinic of Auxologia and Pediatric Endocrinology of the Pediatric Clinic of the Major Hospital of Charity of Novara, while the examination of the BIA will be carried out at the Endocrinology Clinic of the Major Hospital of Charity of Novara.

EXPECTED RESULTS It is expected a change in the body mass index based on the BMI z-score and an improvement in body composition after 6 months from the first visit and then from the implementation of the dietary scheme. In addition, an improvement in metabolic parameters is expected (insulin resistance, glycidic intolerance, dyslipidemia, hepatic steatosis)

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 17 years;
* BMI compatible with obesity or overweight according to IOTF criteria
* Signature of informed consent by parents/legal tutors.

Exclusion Criteria:

* Age below 6 years or over 18
* Previous diagnosis of diabetes mellitus type 2 already placed in dietary or pharmacological therapy
* Subjects already included in dieto-therapeutic regimen
* Obesity secondary to diseases: genetic (Prader Willi syndrome, Down syndrome); metabolic and endocrine (Cushing syndrome, hypothyroidism)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 6-17 years pediatric subjects with obesity or overweight
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Body composition | Change of body composition at baseline (V0) and after 3 months (V3) and 6 months (V6)
  evaluation of body composition with Bioimpendence analysis (BIA)

SECONDARY OUTCOMES:
Dietary compliance with questionnaires | Change of dietary compliance at baseline (V0) and after 3 months (V3) and 6 months (V6)
  Assessment of food conformity, in particular adherence to the Mediterranean diet, through KIDMED questionnaires. The questionnaire will provide a value equivalent to + or - 1 depending on the positive (+1) or negative (-1) response to the questions. Adding up the values will give a final result from which to determine if the current diet is Mediterranean or very different. The scale of values is as follows: less than or equal to 3 indicates a low adhesion, between 4 and 7 an average adhesion and higher than 8 a high adherence to a Mediterranean diet.
Correlation between change in body composition (primary outcome) and dietary compliance (secondary outcome) | Change of dietary compliance at baseline (V0) and after 3 months (V3) and 6 months (V6). Change of BMI at baseline (V0) and after 3 months (V3) and 6 months (V6)
  Subsequent correlation with the primary objective, so with the body composition measured through the analysis of bioimpedance. Observation between the adherence to the diet and the change in body composition, measured through the BIA analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Simonetta Bellone, MD, Principal Investigator — AOU Maggiore della Carità
Locations (1):
- SCDU Pediatria, AOU Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grosso G, Marventano S, Yang J, Micek A, Pajak A, Scalfi L, Galvano F, Kales SN. A comprehensive meta-analysis on evidence of Mediterranean diet and cardiovascular disease: Are individual components equal? Crit Rev Food Sci Nutr. 2017 Oct 13;57(15):3218-3232. doi: 10.1080/10408398.2015.1107021. PMID 26528631
- [Background] Tremmel M, Gerdtham UG, Nilsson PM, Saha S. Economic Burden of Obesity: A Systematic Literature Review. Int J Environ Res Public Health. 2017 Apr 19;14(4):435. doi: 10.3390/ijerph14040435. PMID 28422077
- [Background] Valerio G, Maffeis C, Saggese G, Ambruzzi MA, Balsamo A, Bellone S, Bergamini M, Bernasconi S, Bona G, Calcaterra V, Canali T, Caroli M, Chiarelli F, Corciulo N, Crino A, Di Bonito P, Di Pietrantonio V, Di Pietro M, Di Sessa A, Diamanti A, Doria M, Fintini D, Franceschi R, Franzese A, Giussani M, Grugni G, Iafusco D, Iughetti L, Lamborghini A, Licenziati MR, Limauro R, Maltoni G, Manco M, Reggiani LM, Marcovecchio L, Marsciani A, Del Giudice EM, Morandi A, Morino G, Moro B, Nobili V, Perrone L, Picca M, Pietrobelli A, Privitera F, Purromuto S, Ragusa L, Ricotti R, Santamaria F, Sartori C, Stilli S, Street ME, Tanas R, Trifiro G, Umano GR, Vania A, Verduci E, Zito E. Diagnosis, treatment and prevention of pediatric obesity: consensus position statement of the Italian Society for Pediatric Endocrinology and Diabetology and the Italian Society of Pediatrics. Ital J Pediatr. 2018 Jul 31;44(1):88. doi: 10.1186/s13052-018-0525-6. PMID 30064525
- [Background] Khalil SF, Mohktar MS, Ibrahim F. The theory and fundamentals of bioimpedance analysis in clinical status monitoring and diagnosis of diseases. Sensors (Basel). 2014 Jun 19;14(6):10895-928. doi: 10.3390/s140610895. PMID 24949644
- [Background] Cacciari E, Milani S, Balsamo A, Spada E, Bona G, Cavallo L, Cerutti F, Gargantini L, Greggio N, Tonini G, Cicognani A. Italian cross-sectional growth charts for height, weight and BMI (2 to 20 yr). J Endocrinol Invest. 2006 Jul-Aug;29(7):581-93. doi: 10.1007/BF03344156. PMID 16957405
- [Background] Serra-Majem L, Ribas L, Ngo J, Ortega RM, Garcia A, Perez-Rodrigo C, Aranceta J. Food, youth and the Mediterranean diet in Spain. Development of KIDMED, Mediterranean Diet Quality Index in children and adolescents. Public Health Nutr. 2004 Oct;7(7):931-5. doi: 10.1079/phn2004556. PMID 15482620
- [Background] Hagstromer M, Bergman P, De Bourdeaudhuij I, Ortega FB, Ruiz JR, Manios Y, Rey-Lopez JP, Phillipp K, von Berlepsch J, Sjostrom M; HELENA Study Group. Concurrent validity of a modified version of the International Physical Activity Questionnaire (IPAQ-A) in European adolescents: The HELENA Study. Int J Obes (Lond). 2008 Nov;32 Suppl 5:S42-8. doi: 10.1038/ijo.2008.182. PMID 19011653
- [Background] Chen PS, Chang KC, Chang CH, Chen YT, Huang HW, Tsai SM, Yang HR, Tung YC, Wu WW, Chen HL. The effect of a multidisciplinary lifestyle modification program for obese and overweight children. J Formos Med Assoc. 2022 Sep;121(9):1773-1785. doi: 10.1016/j.jfma.2022.01.011. Epub 2022 Jan 29. PMID 35094911
- See also: Okkio alla salute Data — https://www.epicentro.iss.it/okkioallasalute/indagine-2019-dati

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT06312280/Prot_SAP_000.pdf